CLINICAL TRIAL: NCT05421078
Title: A Placebo-Controlled, Double-Blind, Randomized, Phase 2 Dose-Finding Study to Evaluate the Effect of Obicetrapib as an Adjunct to Stable Statin Therapy in Japanese Subjects.
Brief Title: A Dose-Finding Study in Japanese Patients to Evaluate the Effect of Obicetrapib as an Adjunct to Stable Statin Therapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-8995-203
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-09

CONDITIONS: Dyslipidemia; Hypercholesterolemia; High Cholesterol
Keywords: obicetrapib; statin; LDL-C cholestero; l atherosclerosis
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blind, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo tablet made to resemble active product
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (Placebo Comparator): Once-daily placebo
  Interventions: Drug: Placebo
- 2.5 mg Obicetrapib (Experimental): once-daily Obicetrapib
  Interventions: Drug: Obicetrapib
- 5 mg Obicetrapib (Experimental): once-daily Obicetrapib
  Interventions: Drug: Obicetrapib
- 10 mg Obicetrapib (Experimental): once-daily Obicetrapib
  Interventions: Drug: Obicetrapib

INTERVENTIONS:
Drug: Obicetrapib — tablet
  Other Names: CETP inhibitor
  Arms: 10 mg Obicetrapib; 2.5 mg Obicetrapib; 5 mg Obicetrapib
Drug: Placebo — No active ingredient
  Other Names: placebo tablet
  Arms: Placebo

SUMMARY:
This study will be a placebo-controlled, double-blind, randomized, phase 2 dose-finding study in Japanese patients to evaluate the efficacy, safety, and tolerability of obicetrapib as an adjunct to stable statin therapy.

DETAILED DESCRIPTION:
This study will be a placebo-controlled, double-blind, randomized, phase 2 dose-finding study to evaluate the efficacy, safety, and tolerability of obicetrapib as an adjunct to stable statin therapy in Japanese patients. The screening period for this study will take up to 2-weeks. Afterwards, patients will be randomized to placebo, 2.5 mg obicetrapib, 5 mg obicetrapib or 10 mg obicetrapib for an 8-week treatment period. After the treatment period, patients will continue for a 4-week safety follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C > 70 mg/dL and TG < 400 mg/dL,
* Treated with a stable statin therapy; Atorvastatin 20/40 or Simvastatin 10/20

Exclusion Criteria:

* BMI > or =35 kg/m2
* Significant cardiovascular disease
* HbA1c > 10%
* Uncontrolled hypertension
* Active muscle disease
* GFR < 60 ml/min
* Hepatic dysfunction
* Anemia
* Existing CETP deficiency
* History of Homozygous Familial Hypercholerstrolemia
* History of malignancy
* Alcohol abuse
* Treatment with investigational product
* Treatment with PCSK9
* Clinically significant condition
* Known CETP inhibitor allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ditmarsch, MD, Study Director — NewAmsterdam Pharma
Locations (10):
- Japan (10):
  - Nippon Kokan Fukuyama Hospital, Fukuyama
  - Nakamura Cardiology and Cardiovascular Surgery Clinic, Itoshima
  - Kishiwada Tokushu-Kai Hospital, Osaka
  - Kyosokai AMC NISHI-UMEDA Clinic, Osaka
  - Sakurabashi Watanabe Hospital, Osaka
  - Uji Tokushu-Kai Hospital, Osaka
  - Sanai Hospital, Saitama
  - Shinden Higashi Clinic, Sendai
  - Soka-Sugiura Clinic, Sōka
  - Sugiura Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Once-daily placebo
  Obicetrapib: No active ingredient
- Experimental 2.5 mg Obicetrapib; Experimental 5 mg Obicetrapib; Experimental 10 mg Obicetrapib: once-daily Obicetrapib
  Obicetrapib: tablet
Period: Overall Study
Arm/Group | Placebo | Experimental 2.5 mg Obicetrapib | Experimental 5 mg Obicetrapib | Experimental 10 mg Obicetrapib
Started | 26 | 25 | 25 | 26
Completed | 26 | 25 | 25 | 26
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Population is defined as all participants who received at least one dose of study drug and had a baseline value for LDL-C assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib | Total
Number analyzed (Participants) | 26 | 25 | 25 | 26 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (9.44) | 65.8 (8.09) | 67.8 (9.46) | 62.5 (9.90) | 64.8 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 6 | 7 | 29
  Male | 20 | 15 | 19 | 19 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 25 | 25 | 26 | 102
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 26 | 25 | 25 | 26 | 102
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline Low-Density Lipoprotein Cholesterol (LDL-C) Values [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Measure Description: Baseline LDL-C is defined as the last measurement prior to the first dose of study drug. LDL-C was calculated using the Friedewald Formula.
  milligrams per deciliter (mg/dL) | 110.1 (37.13) | 102.2 (26.58) | 106.4 (27.54) | 109.1 (32.47) | 106.95 (30.93)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) [Friedewald]
Description: Mean percent change from Day 1 to Day 56 in Low-Density Lipoprotein Cholesterol (LDL-C) for each obicetrapib group compared to the placebo group. LDL-C was calculated using the Friedewald equation unless TG≥400 mg/dL or LDL-C ≤50 mg/dL; if TG ≥400 mg/dL or LDL-C ≤50 mg/dL, then LDL-C level was measured directly by preparative ultracentrifugation (PUC).
Time Frame: 8 Weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | -0.78 (14.581) | -25.90 (21.259) | -33.78 (13.247) | -36.80 (25.727)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -25.84, 95% CI 2-sided [-36.53 to -15.14], Standard Error of Mean 5.387
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -33.34, 95% CI 2-sided [-44.01 to -22.66], Standard Error of Mean 5.378
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -36.12, 95% CI 2-sided [-46.68 to -25.55], Standard Error of Mean 5.323

2. Primary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) [Friedewald]
Description: Median percent change from Day 1 to Day 56 in Low-Density Lipoprotein Cholesterol (LDL-C) for each obicetrapib group compared to the placebo group. LDL-C was calculated using the Friedewald equation unless TG≥400 mg/dL or LDL-C ≤50 mg/dL; if TG ≥400 mg/dL or LDL-C ≤50 mg/dL, then LDL-C level was measured directly by preparative ultracentrifugation (PUC).
Time Frame: 8 Weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | -0.89 [-38.6 to 27.8] | -24.81 [-66.0 to 17.7] | -31.94 [-56.8 to -2.9] | -45.80 [-73.0 to 45.5]
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; p value is calculated; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -25.84, 95% CI 2-sided [-36.53 to -15.14], Standard Error of Mean 5.387
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -33.34, 95% CI 2-sided [-44.01 to -22.66], Standard Error of Mean 5.378
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -36.12, 95% CI 2-sided [-46.68 to -25.55], Standard Error of Mean 5.323

3. Primary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) [Friedewald]
Description: LS Mean percent change from Day 1 to Day 56 in Low-Density Lipoprotein Cholesterol (LDL-C) for each obicetrapib group compared to the placebo group. LDL-C was calculated using the Friedewald equation unless TG≥400 mg/dL or LDL-C ≤50 mg/dL; if TG ≥400 mg/dL or LDL-C ≤50 mg/dL, then LDL-C level was measured directly by preparative ultracentrifugation (PUC).
Time Frame: 8 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | -0.48 (3.766) | -26.32 (3.844) | -33.82 (3.838) | -36.60 (3.765)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -25.84, 95% CI 2-sided [-36.53 to -15.14], Standard Error of Mean 5.387
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -33.34, 95% CI 2-sided [-44.01 to -22.66], Standard Error of Mean 5.378
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -36.12, 95% CI 2-sided [-46.68 to -25.55], Standard Error of Mean 5.323

4. Primary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) [PUC]
Description: Mean Percent change from Day 1 to Day 56 in Low-Density Lipoprotein Cholesterol (LDL-C) for each obicetrapib group compared to the placebo group. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 8 Weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | 0.43 (15.456) | -26.10 (23.477) | -30.50 (14.959) | -36.29 (24.513)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; Test type: Superiority; p < .0001, ANCOVA — p value is calculated; Least Squares (LS) Means = -27.20, 95% CI 2-sided [-38.37 to -16.04], Standard Error of Mean 5.626
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, ANCOVA — p value is calculated; Least Squares (LS) Means = -31.23, 95% CI 2-sided [-42.36 to -20.10], Standard Error of Mean 5.609
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, ANCOVA — p value is calculated; Least Squares (LS) Means = -36.81, 95% CI 2-sided [-47.83 to -25.80], Standard Error of Mean 5.550

5. Primary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) [PUC]
Description: Median Percent change from Day 1 to Day 56 in Low-Density Lipoprotein Cholesterol (LDL-C) for each obicetrapib group compared to the placebo group. LDL-C level was measured by preparative ultracentrifugation (PUC)
Time Frame: 8 Weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | 0.67 [-35.3 to 32.5] | -25.97 [-67.6 to 41.9] | -30.40 [-57.8 to -2.7] | -43.72 [-72.0 to 30.9]
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; Test type: Superiority; p < .0001, ANCOVA — p value is calculated; Least Squares (LS) Means = -27.20, 95% CI 2-sided [-38.37 to -16.04], Standard Error of Mean 5.626
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, ANCOVA — p value is calculated; Least Squares (LS) Means = -31.23, 95% CI 2-sided [-42.36 to -20.10], Standard Error of Mean 5.609
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, ANCOVA — p value is calculated; Least Squares (LS) Means = -36.81, 95% CI 2-sided [-47.83 to -25.80], Standard Error of Mean 5.550

6. Primary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) [PUC]
Description: as for outcome 4
Time Frame: 8 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | 0.69 (3.928) | -26.51 (4.013) | -30.54 (4.002) | -36.12 (3.926)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; Test type: Superiority; p < .0001, ANCOVA — p value is calculated; Least Squares (LS) Means = -27.20, 95% CI 2-sided [-38.37 to -16.04], Standard Error of Mean 5.626
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, ANCOVA — p value is calculated; Least Squares (LS) Means = -31.23, 95% CI 2-sided [-42.36 to -20.10], Standard Error of Mean 5.609
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, ANCOVA — p value is calculated; Least Squares (LS) Means = -36.81, 95% CI 2-sided [-47.83 to -25.80], Standard Error of Mean 5.550

7. Secondary Outcome: Mean Percent Change in Apolipoprotein B (ApoB)
Description: Mean percent change from baseline to Day 56 in apolipoprotein B (ApoB) (mg/dL) for each obicetrapib group compared with the placebo group.
Time Frame: 8 Weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | -1.23 (10.614) | -19.80 (15.363) | -24.48 (13.909) | -26.66 (15.0)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -19.00, 95% CI 2-sided [-25.83 to -12.18], Standard Error of Mean 3.439
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -22.45, 95% CI 2-sided [-29.28 to -15.62], Standard Error of Mean 3.441
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -24.86, 95% CI 2-sided [-31.62 to -18.10], Standard Error of Mean 3.406

8. Secondary Outcome: Median Percent Change in Apolipoprotein B (ApoB)
Description: Median percent change from baseline to Day 56 in apolipoprotein B (ApoB) (mg/dL) for each obicetrapib group compared with the placebo group.
Time Frame: 8 Weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | -0.36 [-26.1 to 21.7] | -22.50 [-45.6 to 12.7] | -21.43 [-53.4 to 1.0] | -29.67 [-56.4 to 9.5]
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -19.00, 95% CI 2-sided [-25.83 to -12.18], Standard Error of Mean 3.439
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -22.45, 95% CI 2-sided [-29.28 to -15.62], Standard Error of Mean 3.441
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -24.86, 95% CI 2-sided [-31.62 to -18.10], Standard Error of Mean 3.406

9. Secondary Outcome: LS Mean Percent Change in Apolipoprotein B (ApoB)
Description: as for outcome 8
Time Frame: 8 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | -1.42 (2.407) | -20.43 (2.457) | -23.87 (2.457) | -26.29 (2.408)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -19.00, 95% CI 2-sided [-25.83 to -12.18], Standard Error of Mean 3.439
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -22.45, 95% CI 2-sided [-29.28 to -15.62], Standard Error of Mean 3.441
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -24.86, 95% CI 2-sided [-31.62 to -18.10], Standard Error of Mean 3.406

10. Secondary Outcome: Mean Percent Change in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: Mean percent change from baseline to Day 56 in non-high-density lipoprotein cholesterol (non-HDL-C) (mg/dL) for each obicetrapib group compared with the placebo group
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | -1.80 (12.328) | -25.42 (19.280) | -30.38 (13.839) | -30.25 (23.318)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; Least Squares (LS) Means = -23.94, 95% CI 2-sided [-33.56 to -14.31], Standard Error of Mean 4.850
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -28.39, 95% CI 2-sided [-38.01 to -18.76], Standard Error of Mean 4.849
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -28.55, 95% CI 2-sided [-38.08 to -19.03], Standard Error of Mean 4.801

11. Secondary Outcome: Median Percent Change in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: Median percent change from baseline to Day 56 in non-high-density lipoprotein cholesterol (non-HDL-C) (mg/dL) for each obicetrapib group compared with the placebo group
Time Frame: 8 Weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | -0.37 [-33.3 to 24.2] | -23.74 [-62.4 to 15.6] | -29.82 [-52.8 to 1.3] | -36.96 [-66.3 to 35.8]
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -23.94, 95% CI 2-sided [-33.56 to -14.31], Standard Error of Mean 4.850
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -28.39, 95% CI 2-sided [-38.01 to -18.76], Standard Error of Mean 4.849
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -28.55, 95% CI 2-sided [-38.08 to -19.03], Standard Error of Mean 4.801

12. Secondary Outcome: LS Mean Percent Change in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: LS Mean percent change from baseline to Day 56 in non-high-density lipoprotein cholesterol (non-HDL-C) (mg/dL) for each obicetrapib group compared with the placebo group
Time Frame: 8 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | -1.72 (3.395) | -25.66 (3.463) | -30.11 (3.463) | -30.28 (3.395)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -23.94, 95% CI 2-sided [-33.56 to -14.31], Standard Error of Mean 4.850
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -28.39, 95% CI 2-sided [-38.01 to -18.76], Standard Error of Mean 4.849
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -28.55, 95% CI 2-sided [-38.08 to -19.03], Standard Error of Mean 4.801

13. Secondary Outcome: Mean Percent Change in High-density Lipoprotein Cholesterol (HDL-C)
Description: Mean percent change from baseline to Day 56 in High-density lipoprotein cholesterol (HDL-C) (mg/dL) for each obicetrapib group compared with the placebo group
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | 5.57 (13.271) | 134.75 (56.543) | 153.16 (46.879) | 158.75 (43.171)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 133.11, 95% CI 2-sided [112.85 to 153.36], Standard Error of Mean 10.205
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 147.41, 95% CI 2-sided [127.17 to 167.64], Standard Error of Mean 10.195
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 155.98, 95% CI 2-sided [135.93 to 176.02], Standard Error of Mean 10.100

14. Secondary Outcome: Median Percent Change in High-density Lipoprotein Cholesterol (HDL-C)
Description: Median percent change from baseline to Day 56 in High-density lipoprotein cholesterol (HDL-C) (mg/dL) for each obicetrapib group compared with the placebo group
Time Frame: 8 Weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | 5.22 [-20.7 to 33.3] | 114.29 [57.3 to 307.0] | 144.44 [74.1 to 255.2] | 158.90 [76.6 to 281.6]
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 133.11, 95% CI 2-sided [112.85 to 153.36], Standard Error of Mean 10.205
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 147.41, 95% CI 2-sided [127.17 to 167.64], Standard Error of Mean 10.195
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 155.98, 95% CI 2-sided [135.93 to 176.02], Standard Error of Mean 10.100

15. Secondary Outcome: LS Mean Percent Change in High-density Lipoprotein Cholesterol (HDL-C)
Description: LS Mean percent change from baseline to Day 56 in High-density lipoprotein cholesterol (HDL-C) (mg/dL) for each obicetrapib group compared with the placebo group.
Time Frame: 8 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | 2.5 mg Obicetrapib | 5 mg Obicetrapib | 10 mg Obicetrapib
Number analyzed (Participants) | 26 | 25 | 25 | 26
percent change from baseline | 3.90 (7.141) | 137.00 (7.284) | 151.30 (7.282) | 159.87 (7.139)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 133.11, 95% CI 2-sided [112.85 to 153.36], Standard Error of Mean 10.205
Statistical Analysis 2: Comparison: Placebo vs 5 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 147.41, 95% CI 2-sided [127.17 to 167.64], Standard Error of Mean 10.195
Statistical Analysis 3: Comparison: Placebo vs 10 mg Obicetrapib; Test type: Superiority; p < .0001, Mixed Models Analysis — p value is calculated; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 155.98, 95% CI 2-sided [135.93 to 176.02], Standard Error of Mean 10.100

ADVERSE EVENTS:
Time Frame: From first dose of study drug through Week 12
Description: Safety Population included all participants who received at least 1 dose of any study drug.
Arm/Group | Placebo | Experimental 2.5 mg Obicetrapib | Experimental 5 mg Obicetrapib | Experimental 10 mg Obicetrapib
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 1/25 | 0/26
Other Adverse Events (participants affected / at risk) | 15/26 | 9/25 | 7/25 | 15/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | Experimental 2.5 mg Obicetrapib (N=25) | Experimental 5 mg Obicetrapib (N=25) | Experimental 10 mg Obicetrapib (N=26)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | Experimental 2.5 mg Obicetrapib (N=25) | Experimental 5 mg Obicetrapib (N=25) | Experimental 10 mg Obicetrapib (N=26)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or 12 months after completion of the study, whichever occurs first, Institution may publish the results of its study data. Institution and PI shall provide sponsor with an advance copy of any proposed communications at least 60 days prior and Sponsor shall have 60 days to review. Sponsor may request (a) the deletion of any Confidential Information, (b) reasonable changes, or (c) a delay for an additional period, not to exceed 90 days.

DOCUMENTS (2):
  • Study Protocol (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT05421078/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT05421078/SAP_001.pdf